CLINICAL TRIAL: NCT05171582
Title: The Effect of Periimplantitis Surgical Regenerative Therapy Using Bovine Bone Substitute With Hyaluronic Acid: Randomized Controlled Clinical Trials
Brief Title: Peri-implantitis Surgical Regenerative Therapy Using Bovine Bone Substitute With Hyaluronic Acid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Botiss Medical AG (Other)
Collaborators: Military Medical Academy, Bulgaria (Other)
Responsible Party: Principal Investigator, Dragana Rakasevic, Principal Investigator and Research Associate, Botiss Medical AG
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36/25
Record Dates: First submitted 2021-12-12; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Peri-Implantitis
Keywords: regenerative surgery, periimplantitis, photodynamic therapy
MeSH Terms: conditions — Peri-Implantitis | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Masking Description: Single Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery 1 (Test group) (Active Comparator): In the test group (T), bone defects will be full-filled with bovine bone substitute with HA (Cerabone plus, Botiss, Germany)
  Interventions: Procedure: Surgery 1 (Test group)
- Surgery 2 (Control group) (Active Comparator): In the control group (C), bone defects will be full-filled with xenograft bovine bone substitute without HA (Cerabone, Botiss, Germany).
  Interventions: Procedure: Surgery 2 (Control group)

INTERVENTIONS:
Procedure: Surgery 1 (Test group) — After local anaesthesia, a full-mucoperiosteal flap will be evaluated. After granulation tissue is removed by using titanium or graphite curettes and implant surface decontamination will be performed using photodynamic therapy. Thereafter, the peri-implant bone defects in the test group will be full-filled either with bovine bone substitute with hyaluronic acid (Cerabone plus). Collagen dermal matrix (Mucoderm) will be inserted instead of a collagen membrane. Mucoderm will be fixed with 5.0 resorbable sutures. The flap will be coronally positioned and sutured with 5.0 non-resorbable sutures, respectively.
  Arms: Surgery 1 (Test group)
Procedure: Surgery 2 (Control group) — After local anaesthesia, a full-mucoperiosteal flap will be evaluated. After granulation tissue is removed by using titanium or graphite curettes and implant surface decontamination will be performed using photodynamic therapy. Thereafter, the peri-implant bone defects in the control group will be full-filled either with bovine bone substitute (Cerabone). Collagen dermal matrix (Mucoderm) will be inserted instead of a collagen membrane. Mucoderm will be fixed with 5.0 resorbable sutures. The flap will be coronally positioned and sutured with 5.0 non-resorbable sutures, respectively.
  Arms: Surgery 2 (Control group)

SUMMARY:
The study aimed to assess 6- and 12-months evaluation of clinical, microbiological, and radiography outcomes after performing peri-implantitis regenerative surgical therapy with the bovine bone substitute with or without hyaluronic acid.

Materials and Methods: The study could be designed as randomized control clinical trial. Patients with a minimum of one or more early, moderate and advanced stages of the peri-implant lesion will be included in the study. After meeting inclusion criteria, during a regenerative surgical procedure, after mucoperiosteal flap elevation and implant surface decontamination, all patients will be randomly divided into two groups: test group in which bovine bone substitute with hyaluronic acid (HA) (Cerabone plus, Botiss, Germany) will be applied for the filling peri-implant bone defects while in the control group peri-implant bone defects will be filled with bovine bone substitute (Cerabone, Botiss, Germany). Bone grafts will be covered in both groups with collagen dermal matrix (Mucoderm, Botiss, Germany). Clinical, radiograph and microbiological outcomes will be followed at 6 and 12 months after the surgical procedure. ISQ implant stability will be measured before, during a surgical procedure, and 7, 15, 30 days, 3, 6 and 12 months after a surgical procedure.

DETAILED DESCRIPTION:
Treatment procedure

After the crown was removed immediately, ISQ implant stability and clinical parameters will be measured, and the sample for microbiological analyses will be taken.

Subsequently, patients with a minimum of one or more diagnosed periimplantitis will undergo non-surgical periimplantitis therapy in order to reduce inflammation. The patient will be instructed on adequate oral hygiene. Antibiotics and mouths wash will not be prescribed in this phase.

Surgical procedure

Two weeks after the non-surgical procedure, surgical regenerative therapy will be performed by experienced operators. After local anaesthesia, a full-mucoperiosteal flap will be evaluated. ISQ implant stability will be measured before implant debridement. After granulation tissue is removed by using titanium or graphite curettes, ISQ implant stability will be measured, and implant surface decontamination will be performed, respectively. Implant surface decontamination will be performed by titanium brushes and photodynamic therapy. After implant surface decontamination, bone defect and soft tissue thickness will be measured intra-operatively using a periodontal probe. In the cases where there is additional supracrestal bone lost the implantoplasty will be performed. Thereafter, the bone defects around treated implants will be full-filled either with bovine bone substitute with or without HA (Cerabone plus or Cerabone) and Mucoderm will be inserted. Microderm (Botiss, Germany) will be fixed with 5.0 resorbable sutures. The flap will be coronally positioned and sutured with 5.0 non-resorbable sutures, respectively.

ISQ implant stability will be measured after the flap was sutured. The temporary crown will be inserted, respectively.

Patients will be prescribed antibiotics (Amoxicillin 500 mg, three times per day, in seven days), and 0,12% chlorhexidine solution for 14 days. Sutures will be removed 7 days after surgery.

Prosthetic outcomes

Every patient with periimplantitis will be scanned with an intraoral scanner in order to define premature contacts or interferent contacts in excentre movements of implants. The scan will be taken before any therapy, six, and 12 months after the surgical therapy.

In the first visit, where it is possible, the crown will be removed, and the impression for the temporary crown will be taken, depending on group distribution. A temporary crown will be fixed immediately after the surgical procedure, while the new permanent crown will be made a minimum of three months after surgery. Crowns will be screw-retained. Dental implant emergent profile will be evaluated at 6 and 12 months after prosthetic rehabilitation.

Gained results will be statistically analyzed using SPSS softer.

ELIGIBILITY:
Inclusion Criteria:

Peri-implantitis with:

1. Presence of peri-implant pocket > 5mm,
2. Bleeding on probing (BOP),
3. Radiographic evidence of bone loss > 3mm, or one or two-third bone loss
4. Implant in function for more than one year (prosthetic rehabilitation for more than six months)
5. Good level of oral hygiene (plaque index <1)
6. No periodontal or peri-implant treatment three months prior to the study
7. No use antibiotics in the last three months
8. No anti-inflammatory drugs were used in the previous two months

Exclusion Criteria:

* Buccally implant placement, implant mobility, two-third of bone loss, patient with systemic conditions (diabetes mellitus, leukemia), patient on radiation therapy, drug and alcohol abuse, pregnant and breastfeeding, women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 1. >18 years of age
  2. Competent to fully understand all information regarding the research protocol of the study and to sign a written consent for participation
Enrollment: 25 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
Change of clinical attachment level (CAL) | Change from baseline CAL at 12 months
  CAL, measured in millimetres as the distance from implant shoulder to the bottom of peri-implant pocket at six points.
Change of Peri-implant probing depths (PPD) | Change from baseline PPD at 12 months
  PPD, measured in millimetres as the distance from mucosal margin to bottom of periodontal pocket.

SECONDARY OUTCOMES:
Change of Keratinized tissue width (KTW) | Change from baseline KTW at 12 months
  KTW, measured at the middle of the inserted implant in the millimetres as the distance between MM of the implant to a mucogingival junction (MGJ).
Change of gingival thickness (GT) | Change from baseline GT at 12 months
  GT, measured at the mid-buccal aspect of treated implants on the long axis, 3 mm apically from perimucosal tissue margin.
Healing index (HI) score | Changes of the wound healing within 30 days
  Assess of the wound healing based on redness, granulation tissue presence, bleeding, suppuration, and epithelialization

OTHER OUTCOMES:
Radiography measurements of peri-implant defects | Measured at baseline and 12 months
  Radiography measurements of peri-implant defects will be performed using CBCT and x-ray

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dental Medicine, University of Belgrade, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Will be published in International Journal
Supporting Information: Study Protocol, CSR
Time Frame: from 2022. to 2024.
Access Criteria: There are no access criteria

REFERENCES:
- [Background] Albrektsson T, Canullo L, Cochran D, De Bruyn H. "Peri-Implantitis": A Complication of a Foreign Body or a Man-Made "Disease". Facts and Fiction. Clin Implant Dent Relat Res. 2016 Aug;18(4):840-9. doi: 10.1111/cid.12427. Epub 2016 May 30. PMID 27238274
- [Background] Mombelli A. Etiology, diagnosis, and treatment considerations in peri-implantitis. Curr Opin Periodontol. 1997;4:127-36. PMID 9655032
- [Background] Schwarz F, Jepsen S, Herten M, Sager M, Rothamel D, Becker J. Influence of different treatment approaches on non-submerged and submerged healing of ligature induced peri-implantitis lesions: an experimental study in dogs. J Clin Periodontol. 2006 Aug;33(8):584-95. doi: 10.1111/j.1600-051X.2006.00956.x. PMID 16899102
- [Background] Schwarz F, Sahm N, Bieling K, Becker J. Surgical regenerative treatment of peri-implantitis lesions using a nanocrystalline hydroxyapatite or a natural bone mineral in combination with a collagen membrane: a four-year clinical follow-up report. J Clin Periodontol. 2009 Sep;36(9):807-14. doi: 10.1111/j.1600-051X.2009.01443.x. Epub 2009 Jul 21. PMID 19637997
- [Result] Schwarz F, Derks J, Monje A, Wang HL. Peri-implantitis. J Periodontol. 2018 Jun;89 Suppl 1:S267-S290. doi: 10.1002/JPER.16-0350. PMID 29926957